CLINICAL TRIAL: NCT03679169
Title: Randomized Controlled Trial for the Evaluation of Complete Microscopic Resection Margin (R0) and Lymph Node Involvement After Standard Pancreatosplenectomy (SPS) Versus Radical Anterograde Modular Pancreatosplenectomy (RAMPS)
Brief Title: Evaluation of Complete microscopicE Resection Margin (R0) and Lymph Node Involvement After Standard Pancreatosplenectomy (SPS) Versus Radical Anterograde Modular Pancreatosplenectomy
Acronym: REMIND-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REMIND-01-IPC 2017-050
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group RAMPS (Experimental): Radical antegrade modular pancreatosplenectomy
  Interventions: Procedure: pancreatosplenectomy
- Group SPS (Active Comparator): standard pancreatosplenectomy
  Interventions: Procedure: pancreatosplenectomy

INTERVENTIONS:
Procedure: pancreatosplenectomy — standard or radical anterograde modularpancreatosplenectomy

SUMMARY:
Resection with negative margins (R0) followed by adjuvant chemotherapy is today the standard of care and the only chance of cure for patients with pancreatic ductal adenocarcinoma (PDA). Incomplete microscopic resection margin (R1) after pancreatic resection has been reported to occur in 17 to >80% of cases depending on the nonconsensual definition of R1 status. This discrepancy is reflected in conflicting reports regarding the prognostic relevance of R1 resection. Currently, neither the definition of the margin involvement nor the surgical technique to clear the margins is consistently applied, resulting in conflicting data in the literature. The Radical Antegrade Modular Pancreatosplenectomy (RAMPS) was described by Strasberg et al. in 2003 to increase the rate of R0 resection for left PDA. However, there is no grade A recommendation and surgical practices still remain heterogeneous as many surgeons still consider the "retrograde" technique as the standard procedure. The invasion of the resection margins is often poorly evaluated, including in large clinical trials. The surgical specimens are not systematically inked and the microscopic invasion of the splenic vessels is underreported, leading to inaccurate pathologic evaluation.

A French prospective multicenter study (Delpero JR et al; ClinicalTrials.gov: NCT00918853) was previously conducted for pancreaticoduodenectomy specimens. A recent update (Ann Surg 2017, in press) has emphasized the value of a standardized pathology protocol to accurately assess the impact of R0 resection and improve patient's stratification.

Today, no recommendations are available regarding the surgical procedure and histological analysis for DP specimen handling.

The primary endpoint of this multicenter randomized control trial (RCT) is to investigate the benefit of the RAMPS procedure in comparison to standard distal pancreatosplenectomy (SDPS) on the R0-resection rate using a high-quality pathology protocol. To date, there are no prospective data assessing the superiority of the RAMPS technique over standard resection. This study will be the first RCT on the subject.

This study could improve the surgical practices and define a surgical standard of care. The pathology protocol used for the study could help to standardize histopathology report on margin status. It could also provide a better evaluation of the impact of adjuvant and neoadjuvant therapies on local control. This study should lead to improved selection of patients for upfront surgery and give appropriate perioperative treatment tailored to a well-defined disease stage. Furthermore, guidelines for surgical practices and standardization of histological examination may represent a significant step forward in the design of future trials to assess perioperative strategies.

DETAILED DESCRIPTION:
Resection with negative margins (R0) followed by adjuvant chemotherapy is today the standard of care and the only chance of cure for patients with pancreatic ductal adenocarcinoma (PDA). For distal pancreatectomy (DP), lymph node disease and R1 resection are mainly underreported owing to the lack of available consensus about the minimum number of lymph nodes to be assessed and the definition of the margin status. Incomplete microscopic resection margin (R1) after pancreatic resection has been reported to occur in 17 to >80% of cases depending on the nonconsensual definition of R1 status. This discrepancy is reflected in conflicting reports regarding the prognostic relevance of R1 resection. Currently, neither the definition of the margin involvement nor the surgical technique to clear the margins is consistently applied, resulting in conflicting data in the literature. The Radical Antegrade Modular Pancreatosplenectomy (RAMPS) was described by Strasberg et al. in 2003 to increase the rate of R0 resection for left PDA. During the procedure the pancreatic transection is performed in front of the mesentericoportal venous axis; the lymphadenectomy extends from the left side of the celiac trunk to the left hemicirconference of the superior mesenteric artery; the anterior renal fascia is removed. However, there is no grade A recommendation and surgical practices still remain heterogeneous as many surgeons still consider the "retrograde" technique as the standard procedure. The invasion of the resection margins is often poorly evaluated, including in large clinical trials. The surgical specimens are not systematically inked and the microscopic invasion of the splenic vessels is underreported, leading to inaccurate pathologic evaluation.

A French prospective multicenter study (Delpero JR et al; ClinicalTrials.gov: NCT00918853) was previously conducted for pancreaticoduodenectomy specimens. A recent update (Ann Surg 2017, in press) has emphasized the value of a standardized pathology protocol to accurately assess the impact of R0 resection and improve patient's stratification.

Today, no recommendations are available regarding the surgical procedure and histological analysis for DP specimen handling.

Patients enrolled in this study will be randomized (standard resection procedure versus the RAMPS technique) in 20 participating centers. Inclusions are planned over a 3 years-period. Margin resection will be assessed using a standardized histopathologic protocol which will involve axial specimen slicing, extensive tissue sampling and multicolor staining. Specimens will be inked systematically in the operative room. Five margins will be studied: the retroperitoneal margin (with the anterior renal fascia in the "RAMPS" group); the celio-mesenteric artery interface; the portal vein groove; the anterior margin; the pancreatic transection margin. Thus, the inking will identify each face of the "circumferential margin". The splenic vessels involvement will be independently identified and analyzed. The distance between tumor cells and each inked margin (ie: the clearance) will be precisely defined from 0 to 2mm with increments of 0.5mm. The invasion of the splenic vessels will be assessed both on the preoperative CT-scan and the specimens. A second centralized histopathological review of the specimens will be performed by a committee of referents pathologists in pancreatic specimens handling.

The primary endpoint of this multicenter randomized control trial (RCT) is to investigate the benefit of the RAMPS procedure in comparison to standard distal pancreatosplenectomy (SDPS) on the R0-resection rate using a high-quality pathology protocol. Secondary outcome measures will be: a) survival (overall, relapse and progression free survival) according to the two surgical techniques; b) evaluation of the independent determinants of post-resection survival: R1 for each margin at each increment; splenic vessels invasion; LN involvement (and LN ratio).

To date, there are no prospective data assessing the superiority of the RAMPS technique over standard resection. This study will be the first RCT on the subject.

This study could improve the surgical practices and define a surgical standard of care. The pathology protocol used for the study could help to standardize histopathology report on margin status. It could also provide a better evaluation of the impact of adjuvant and neoadjuvant therapies on local control. This study should lead to improved selection of patients for upfront surgery and give appropriate perioperative treatment tailored to a well-defined disease stage. Furthermore, guidelines for surgical practices and standardization of histological examination may represent a significant step forward in the design of future trials to assess perioperative strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Tumor of the body or tail of the pancreas compatible with pancreatic ductal adenocarcinoma before surgery
* Intraductal papillary mucinous neoplasms (IPMN) with invasive carcinoma
* Resectable tumor
* Absence of medical contraindication Borderline* resectable tumors with preoperative treatment could be enlisted in the protocol

Exclusion Criteria:

* Patients with legal protection
* Pregnancy
* Preoperative distant metastasis and unresectable tumor (ie tumor interface with the celiac axis and superior mesenteric artery > 180°, aortic involvement or unreconstructible superior mesenteric venous resection due to tumor involvement or occlusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2022-09-17 (Estimated); Study Completion 2024-09-17 (Estimated)

PRIMARY OUTCOMES:
Rate of resection margins involvement and lymph node involvement between RAMPS and SPS performed for pancreatic adenocarcinoma of the body and tail, using a standardized pathology protocol. | Day of surgery (1 day)
  Comparison of the rate of resection margins involvement and lymph node involvement between RAMPS (radical anterograde modular pancreatosplenectomy) and SPS (standard pancreatosplenectomy) performed for pancreatic adenocarcinoma of the body and tail, using a standardized pathology protocol.

CONTACTS AND LOCATIONS:
Overall Officials: DELPERO Jean-Robert, MD, PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- GENRE, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Institut PAOLI-CALMETTES — http://institutpaolicalmettes.fr